CLINICAL TRIAL: NCT05477342
Title: Comparison of the Effect of Board Game and Tobacco Cessation Education on Nicotine Addiction in Adolescent Smokers: a Randomized Controlled Trial.
Brief Title: Reducing Nicotine Addiction in Adolescent Smokers
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ministry of National Education, Turkey (Other Government)
Responsible Party: Principal Investigator, Remziye CAN, Principal Investigator, Ministry of National Education, Turkey
Allocation: Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: MNETurkey
Record Dates: First submitted 2022-04-03; First posted 2022-07-28 (Actual); Last update posted 2022-07-28 (Actual); Status verified 2022-07

CONDITIONS: Nicotine Dependence, Cigarettes; Cessation, Tobacco; Cessation, Smoking; Adolescent Problem Behavior
Keywords: adolescent; board game; change of stage; dependence; gamification; nicotine
MeSH Terms: conditions — Tobacco Use Disorder; Tobacco Use Cessation; Smoking Cessation

STUDY DESIGN:
Intervention Model Description: Transtheoretical Model
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- İntervention 1 (Experimental): Experimental 1 - Board Game Group: Board game group played only board game.
  Interventions: Behavioral: Board Game
- İntervention 2 (Experimental): Experimental 2 - Tobacco Cessation Education Group: The Tobacco Cessation Education Group received only education according to the stages of change model.
  Interventions: Behavioral: Tobacco Cesseation Education
- İntervention 3 (Experimental): Experimental 3 - Combined intervention Group:Combined intervention group received both board game and tobacco cessation education.
  Interventions: Behavioral: Combined İntervention
- Control Group (No Intervention): No intervention was made in the control group.

INTERVENTIONS:
Behavioral: Board Game — The BG group that will play the game were divided into four groups with five or six participants in each group. (GP (Game Player) GP1- GP 2- GP 3- GP 4.
  Arms: İntervention 1
Behavioral: Tobacco Cesseation Education — The TCE group were divided three group that E1 (Precontemplation) -E2 (Contemplation)-E3 (Preparation) according to the thinking stages scale.
  Arms: İntervention 2
Behavioral: Combined İntervention — The CI group was divided into five groups for play that will play the game were divided into four groups with five or six participants in each group. (GP (Game Player)GP 5- GP 6- GP 7- GP 8- GP 9).
  The CI group was divided into three groups for education that E4 (Precontemplation) -E5 (Contemplation)-E6 (Preparation) according to the thinking stages scale.
  Arms: İntervention 3

SUMMARY:
Adolescents are at risk for tobacco use due to factors such as impulsivity, poor perception, desire to prove themselves, and insufficient neurological development. The Center of Disease (CDC) warns that if smoking continues at the current rate among young people, young people younger than 18 will die prematurely from a smoking-related disease

The aim of this study was to comparison the effect of a board game and tobacco cessation education on reducing nicotine addiction in adolescents.

A single-blind randomized controlled trial was used to evaluation the effect s of the different interventions on tobacco cessation. The 12 week interventions included: 1) Board Game (BG) and 2) Tobacco Cessation Education (TCE) developed based on Transtheoretical Model and 3) combined use of these two interventions (Cİ). All interventions were compared to Control Group(CG). "Fagerström Test for Nicotine Dependence (FNTD)" were used to collect data at baseline, at 8.week and at 12.week the intervention. "Assessment Of Stage Of Change Form (ASCF)" were used to collect data at baseline and at the end of each intervention (every two weeks one).

Participants were consisted of students studying at a high school in Eskisehir in Turkey. In order to form the intervention groups, permission was obtained from the school principal and teacher of each class, and the students were informed about the purpose of the study and the participation criteria. It was done in information classes. Recruitment began in October 2018 and end in January 2019.

Students who wanted to participate in the study were asked to send a short message to the investigator's private phone number. An automated response with a hyperlink was sent to a web page where information about the study was presented and students were asked to give informed consent at the push of a button. Students who agreed to participate were enrolled in a web-based questionnaire for egilibility screening.

DETAILED DESCRIPTION:
Tobacco use is one of the leading preventable causes of death.Tobacco use is a major risk factor for cardiovascular and respiratory diseases, more than 20 different types or subtypes of cancer, and many other debilitating health conditions. The risk of morbidity and mortality increases with the increase of tobacco use. There are many methods such as smoking cessation pharmacotherapy, nicotine replacement therapy, cognitive behavioral therapies. One of them is the education aiming at behavior change organized according to the Transtheoretic Model (TTM) . The main purpose of the model is to prevent addiction by applying the change stages without any medical support. However, these techniques have been reported to be limited in quitting success. This situation necessitated the use of different techniques. One of these techniques is games. The game; It is a conscious activity that provides socialization, does not have a specific financial gain/profit purpose, is carried out in a certain time period, according to binding rules, has a special purpose and provides an extraordinary life.Since it is very easy to reach information thanks to technology in our age, teaching activities with traditional methods are boring and cannot provide motivation. Therefore, games can create learning environments that make education fun. While the use of games in health education exposes individuals to subjects, it aims to create an internal motivation, targeting protection and improvement of health.

The sample size of the study was Cohen's effect size calculation. The effect size is generally defined as the size of the difference between the null hypotheses and alternative hypotheses, which is an indicator of the practical significance of the research results. Cohen's effect size calculation varies according to the study design. For our study, the ANOVA effect formula was used which is the intergroup interaction (relationship) test in repeated measurements. For 4 groups and 3 repeated measurements, the total sample size of based on a power of 0.80, with an effect size of 0.175 and a Type I error rate of 0.05 was calculated 80.

Study inclusion criteria were studying at XXX High School, having at least one cigarette a day and volunteering to participate in the study. There were 106 students who smoked regularly every day and were willing to participate in the study. Therefore we calculated the power of study with Type I error rate of 0.05, effect size of 0.175 and 106 samples as 0.91.

For the randomization; after baseline assessment, eligible students was given an automatic number using Java's built-in random number generator and randomly assigned to four equally-probability groups. Randomization was done by a research blind person in the EXCEL program. Research personnel were blind to allocation at initial randomization but were informed after assignment to groups. Participants were informed about which group they were allocated to. There were 26 participants in the BG group, 25 in the TCE group, 26 in the Cİ group, and 26 in the CG.

For the measurements were used Socio-demographic feature identification form,Fagerstrom test for nicotine dependence,Stages of Change Scale.

Socio-demographic feature identification form: The socio-demographic feature identification form prepared by the researcher consisted of questions related to age, gender, class, place of residence, daily cigarette consumption, age of starting smoking, smoking status in parents, and the reason for starting smoking.

Fagerstrom test for nicotine dependence (FTND):It was developed in 1991 by Heatherton et al (Heatherton et al., 1991). The Turkish validity and reliability study of the scale was performed by Uysal et al. in 2003 and its Cronbach's alpha coefficient was found to be 0.56 (Uysal et al., 2004). FTND is a self-assessment scale that provides a Likert-type measurement used to evaluate the risk of nicotine in terms of physical dependence and to measure its level and change in severity.

Stages of Change Scale (SCS): Developed by Prochaska and DiClemente in 1983, SCS shows the stages of change individuals are in when trying to change their problematic behaviors. There is no scoring in the scale. "Have you stopped smoking?" The stage of change is determined according to the answers given by the individual to the question. The response of the individual "I don't plan to quit in the next 6 months" to precontemplation stage , "I intend to quit within 6 months" to contemplation stage, "I intend to quit within 30 days" to preparation stage , "I quit less than 6 months ago" to action stage, "to longer than 6 months" I quit a while ago" indicates that it is in the maintenance stage.

For the interventions; Participants in the TCE and CE groups were splitted three groups, TCE 1 (Precontemplation) -TCE2 (Contemplation)-TCE 3 (Preparation) according to the thinking stages scale. The BG and CI group that will play the game were divided into nine groups with five or six participants in each group. (GP (Game Player) 1- GP 2- GP 3- GP 4- GP 5- GP 6- GP 7- GP 8- GP 9).

Each group (participants in the BG, SA, TCE group) received intervention every two weeks. The Stages of Change Scale (DAS) was administered after each interview. The groups were rearranged before each intervention.

Message groups were created to communicate with the participants. The purpose of creating these message groups was to announce the class and time of each intervention. The interventions were carried out in different classrooms, at different times, by the researcher only, in order to ensure an atmosphere of trust and full benefit from the interventions.

Board Game The Pick-Klop game is a board game played with cards that allows interaction between players. The aim of the game is to help smokers change their attitudes and cognitions about nicotine/cigarette/tobacco addiction. Goals of the game; to inform smokers about tobacco smoking and quitting in a way that does not make them feel guilty, to increase their level of self-confidence in their ability to cessation (self-efficacy), to change attitudes towards tobacco addiction (perceived advantages and disadvantages), and to help people through the cessation process. Cards of game consist of three categories: question card, advantage-disadvantage card, stimulus-punishment card (Khazaal et al., 2008). Question cards are cards that contain questions about tobacco use, its harms, ways to cessation, problems experienced during cessation and ways to cope with these problems. If the player answers correctly in the question category, player gets points same to the number on the dice. Points earned are used in the stimulus-punishment category. Surprise cards are cards that add fun to the game, allowing them to get gifts or hidden cards, help or hinder another player during the game. Stimulus-punishment cards are cards depending on the player's approach, can either cause a return to the starting line of the game or are cards that prevent a return to the beginning by offering alternative behaviors to tobacco smoking behavior.

The game is played with a minimum of two and a maximum of six people. The big dice player starts the game. The game is managed by a moderator who knows the game. The dice are rolled a second time. The pawn is moved by the number on the rolled dice. Whichever category of card is in the box, it draws a card from that category. If the box is in the category of questions, the player who rolls the dice draws a card and gives it to the moderator. The moderator reads the question. İf the player answers the question correctly, gain to points. If the player comes to the surprise card category with the dice roll, chooses from the surprise cards. The player who rolls the dice and falls into the stimulus-punishment card category chooses a card. In the situation indicated on the card, player either says "I smoke" or chooses the strategy to prevent smoking. If the player did not answer the question on the question card correctly or did not choose the anti-smoking strategy on the stimulus-punishment card, they pay points. If player doesn't have enough points, player returns to one of three different levels on the game board. The winning player is the first to reach the final game box. The duration of each game varies between 15-45 minutes, depending on the speed of the player's response and reaching the final game box.

Tobacco Cessation Education Programme The training organized according to the stages of change model was designed by the researchers in the light the Turkish Thoracic Society Smoking Cessation Guide according to the stage of change precontemplation, contemplation, preparation, action, maintenance. TTM was developed by Prochaska and DiClemente in 1982, which is defined as a five-stage process of change: precontemplation, contemplation, preparing, acting, and maintenance, which enables individuals to adapt and determine their readiness for smoking cessation treatment. The model's definition of behavior change as a gradual, continuous and dynamic structure is the most basic feature that distinguishes it from other traditional behaviorist approaches that evaluate behavior change as a sharp and direct result. This model, which was first used in smoking cessation programs, includes sensitive measurement tools that measure the individual's cognitive and behavioral processes, self-confidence about change, perception of decision making and factors that make change difficult. With this feature, it enables the identification of individuals in different stages of behavior change, planning individual-specific interventions, evaluating the effectiveness of implemented interventions and planning new initiatives.

For this study was received approval of the Eskisehir Osmangazi University Clinical Research Ethics Committee (DNR: 80558721/G-313). and Ministry of National Education (DNR: 88074293-605.01-E.3512979.

ELIGIBILITY:
Inclusion Criteria:

* Studying at Odunpazarı Mustafa Kemal Atatürk Vocational and Technical Anatolian High School,
* Having at least one cigarette a day,
* Volunteering to participate in the research

Exclusion Criteria:

* Not smoker
* Not wanting to participate in research
* Have a mental health disorder

Ages: 12 Years to 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 103 (Actual)
Dates: Start 2018-09-03 (Actual); Primary Completion 2018-10-03 (Actual); Study Completion 2018-12-05 (Actual)

PRIMARY OUTCOMES:
Fagerstrom test for nicotine dependence (FTND) | Three month
  The Fagerström Test for Nicotine Dependence is a standard instrument for assessing the that played both the board game and received tobacco cessation education was more successful in education tobacco than the group that played only the board game and received only smoking cessation education.
Stages of Change Scale (SCS): | Three month
  There is no scoring in the scale. "Have you stopped smoking?" The stage of change is determined according to the answers given by the individual to the question. The response of the individual "I don't plan to quit in the next 6 months" to precontemplation stage , "I intend to quit within 6 months" to contemplation stage, "I intend to quit within 30 days" to preparation stage , "I quit less than 6 months ago" to action stage, "to longer than 6 months" I quit a while ago" indicates that it is in the maintenance stage

CONTACTS AND LOCATIONS:
Locations (1):
- Remziye CAN, Tepebaşı, Eski̇şehi̇r, Turkey (Türkiye)